CLINICAL TRIAL: NCT05584683
Title: A Single Dose Study to Determine the Pharmacokinetic Profiles of Amoxicillin and Clavulanate in Pediatric Patients Receiving Either LP-001 or Augmentin ES-600 Orally
Brief Title: A Pharmacokinetic Study of LP-001 in Children With a Bacterial Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kaizen Bioscience Co. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP-001
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Pediatric; Bacterial Infections
Keywords: Amoxicillin; amoxicillin-clavulanate; Clavulanic acid; Bacterial Infections; Anti-Infective Agents
MeSH Terms: conditions — Bacterial Infections | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Intervention Model Description: single site, single dose, open label, pharmacokinetic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LP-001 Arm (Experimental): a novel amoxicillin/clavulanate formulation
  Interventions: Drug: Amoxicillin potassium clavulanate
- Augmentin ES-600 (Active Comparator): Augmentin ES-600
  Interventions: Drug: Amoxicillin potassium clavulanate (Augmentin ES-600)

INTERVENTIONS:
Drug: Amoxicillin potassium clavulanate — LP-001 will be reconstituted and administered as a single dose
  Arms: LP-001 Arm
Drug: Amoxicillin potassium clavulanate (Augmentin ES-600) — Augmentin ES-600 will be reconstituted and administered as a single dose
  Arms: Augmentin ES-600

SUMMARY:
The purpose of this study is to determine the pharmacokinetic profiles of LP-001, an amoxicillin and clavulanate formulation compared to the pharmacokinetic profiles of Augmentin ES-600 for use in pediatric patients with a bacterial infection.

DETAILED DESCRIPTION:
This is a single site, open-label, single dose Phase 1 pharmacokinetic study of LP-001, an amoxicillin and clavulanate formulation, for use in pediatric patients between 3 and 24 months of age with a bacterial infection. 24 pediatric patients will each receive a single dose of LP-001 in a fed state while 15 pediatric patients will each receive a single dose of Augmentin ES-600 in a fed state. 3-4 blood draws per patient will be attempted up to 8 hours post dose.

ELIGIBILITY:
Inclusion Criteria 1. Male or female children who were aged between 3 months and 24 months of age. Patients recruited from urgent care/emergency room or outpatient setting may carry a diagnosis of a mild infection which could include but are not limited to one of the following diagnosis: community acquired pneumonia, aspiration (pneumonia), urinary tract infections, lymphadenitis, retropharyngeal abscess, peritonsillar abscess, animal or human bite, cellulitis, skin abscess, bronchiolitis or dental infection.

2. Since amoxicillin/clavulanic acid is currently only approved for acute otitis media (AOM) by the Food and Drug Administration in the 3-24 month old age range, we will also include a portion of patients recruited from urgent care/emergency room or outpatient setting with a documented AOM diagnosis per provider's exam with planned prescription for amoxicillin or amoxicillin/clavulanic acid to address any of the concerns below: i) onset of symptoms within 48 hours ii) middle ear effusion as demonstrated by ≥2 of the following:

1. decreased or absent mobility of the tympanic membrane
2. yellow or white discoloration of the tympanic membrane
3. opacification of the tympanic membrane. iii) acute inflammation demonstrated by:

(1) moderate or marked bulging of the tympanic membrane, or slight bulging accompanied with apparent otalgia or marked tympanic membrane erythema.

Or A documented OM diagnosis per provider's exam with planned prescription for amoxicillin or amoxicillin/clavulanic acid.

3. Patients recruited from the inpatient setting who have not yet received an amoxicillin containing product (i.e. on an IV antibiotic, or diagnosis and treatment not started until after admission, or diagnosis does not warrant an antibiotic). Examples could include, but are not limited to one of the following diagnosis: acute otitis media, otitis media, community acquired pneumonia, aspiration (pneumonia), urinary tract infections, lymphadenitis, retropharyngeal abscess, peritonsillar abscess, animal or human bite, cellulitis, skin abscess, bronchiolitis or dental infection. If the clinical team decides to transition the patient to an amoxicillin-containing product for continuation of treatment, a single test dose of LP-001 would serve as the first dose of enteral treatment.

4. Written informed consent by the patient's parent or legal guardian and where appropriate.

5. Based upon IRB guidelines, blood volume for PK sampling, based on body weight, will be less than 5% of blood volume per day based upon 70-80 mL blood/kg. Blood sampling will be done between 1-4 time points per patient totaling a blood volume of between 1-3ml.

Exclusion Criteria

Patients will be excluded from the study if they satisfy any of the following criteria:

1. Definite or suspected personal history or family history of significant hypersensitivity, intolerance, or allergy to penicillin, amoxicillin, amoxicillin clavulanate, or aspartame. History of reaction to multiple allergens (if considered clinically relevant by the principal investigator or designee).
2. Children who weigh less than 5 kg or more than 40kg. Patients who are younger than 3 months or older than 24 months (i.e. past their 2nd birthday).
3. Patients with a serious underlying disease, including failure to thrive, which could affect the safety, efficacy, or pharmacokinetics of the study medication.
4. History or presence of gastrointestinal, hepatic, or renal disease or other conditions known to interfere with the absorption, distribution, metabolism or excretion of study medication.
5. History of diarrhea due to Clostridium difficile following treatment with antibiotics.

Have a serious underlying systemic clinical manifestation that may obscure response to infection (eg, cystic fibrosis, neoplasms, or juvenile diabetes), as determined by the investigator (or designee).

7. Have renal or hepatic dysfunction or insufficiency. 8. Have immune dysfunction or are receiving immunosuppressive therapy. 9. Have a chronic gastrointestinal condition (eg, malabsorption or inflammatory bowel disease), as determined by the investigator (or designee).

10. Have phenylketonuria or history of amoxicillin clavulanate associated cholestatic jaundice.

11. Have a systolic blood pressure <60 mmHg or capillary refill >3 seconds. 12. Use of any amoxicillin product within the previous 96 hours. 13. Poor peripheral venous access. 14. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days, current enrollment in another clinical study that could impact the results of this study, or previous enrollment in this clinical study.

15. Patients who, in the opinion of the investigator (or designee), should not participate in this study.

16. Patients related to the sponsor or investigator.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Mean plasma concentration-time curves of amoxicillin and clavulanic acid | 6-8 hours post dose
  Calculation of mean plasma
Area under the serum concentration-time curve (AUC) of amoxicillin and clavulanic acid combination | 6-8 hours post dose
  Calculation of AUC
Maximum serum concentration (Cmax) of amoxicillin and clavulanic acid combination | 6-8 hours post dose
  Calculation of CMAX

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided